CLINICAL TRIAL: NCT01088360
Title: An Observational Cohort to Assess Safety and Outcomes in Patients Treated With Abatacept and Other Anti-Rheumatic Therapies
Brief Title: Safety Study of Abatacept to Treat Rheumatoid Arthritis (B)
Status: Active, not recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: National Data Bank for Rheumatic Diseases (NDB) (Other)
Responsible Party: Sponsor
Other Study IDs: IM101-045B
Record Dates: First submitted 2010-03-12; First posted 2010-03-17 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients with rheumatoid arthritis initiating abatacept
- Pts with RA initiating other biologic disease-modifying drugs
- Pts w/ RA non-biologic disease-modifying anti-rheumatic drugs

SUMMARY:
The purpose of this study is to compare the incidence rates of targeted infections, malignancies and mortality among patients with rheumatoid arthritis who are treated with abatacept and those who are treated with other anti-rheumatic medications.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Diagnosis of rheumatoid arthritis
* > 18 years at index treatment initiation or switch
* Starting treatment with abatacept or new disease-modifying anti-rheumatic drug (including switching or adding) or biologic disease modifying drug.
* Read/write English

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being treated for rheumatoid arthritis in the US
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2005-03-31 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Key safety outcomes (targeted infections, malignancies, mortality) | Every 6 months throughout the study

SECONDARY OUTCOMES:
Patient-reported infusion reactions | Every 6 months throughout the study
Multiple sclerosis, lupus, and psoriasis | Every 6 months throughout the study
Adverse events in pregnant women who receive abatacept | Every 6 months throughout the study
Adverse events in subjects on abatacept who receive concomitant biologics | Every 6 months throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx